CLINICAL TRIAL: NCT02588131
Title: A Single Arm, Phase II Clinical Study of Tremelimumab Combined With the Anti-PD-L1 MEDI4736 Monoclonal Antibody in Unresectable Malignant Mesothelioma Subjects: The NIBIT-MESO-1
Brief Title: A Study of Tremelimumab Combined With the Anti-PD-L1 MEDI4736 Antibody in Malignant Mesothelioma (NIBIT-MESO-1)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Italian Network for Tumor Biotherapy Foundation (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NIBIT-MESO-1
Record Dates: First submitted 2015-10-26; First posted 2015-10-27 (Estimated); Last update posted 2015-10-27 (Estimated); Status verified 2015-10

CONDITIONS: Pleural Mesothelioma; Peritoneal Mesothelioma
Keywords: tremelimumab; anti-PD-L1 MEDI4736 (Durvalumab); malignant mesothelioma
MeSH Terms: conditions — Mesothelioma, Malignant | interventions — tremelimumab; durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- tremelimumab plus MEDI4736 (Experimental): Tremelimumab in combination with MEDI4736
  Interventions: Drug: tremelimumab plus MEDI4736

INTERVENTIONS:
Drug: tremelimumab plus MEDI4736 — tremelimumab1 mg/kg i.v over 60 minutes plus MEDI 4736 20 mg/kg i.v every four weeks for 4 doses, then MEDI4736 20 mg/kg IV every four weeks for additional 9 doses.
  Other Names: MEDI4736 (durvalumab)

SUMMARY:
This phase 2, open-label, single arm study aims to evaluate the efficacy of tremelimumab in combination with the anti-PD-L1 MEDI4736 in patients with unresectable malignant mesothelioma subjects

DETAILED DESCRIPTION:
The prognosis of malignant mesothelioma (MM) patients remains dismal and effective treatment represents a high un-met medical need. Investigators have recently reported promising clinical activity of the anti-CTLA-4 mAb tremelimumab in pre-treated MM patients: disease control rate (DCR) was 31%, and survival rate at 1- and 2-years were 48.3% and 36.7%, respectively. These initial findings were corroborated by a second study in which, based on retrospective pharmacokinetic analyses, an intensified schedule of tremelimumab was utilized. Fifty-two % of patients achieved a DCR (median duration 10.9 months). These intriguing clinical results and the emerging efficacy of immunomodulatory mAb targeting the PD-1/PD-L1 axis in different tumor types, prompted us to design the NIBIT-MESO-1 study aimed to investigate the efficacy of tremelimumab combined with the anti-PD-L1 MEDI4736 in MM patients.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give written informed consent.
* Histologic diagnosis of malignant mesothelioma.
* Subjects who have refused a first line platinum-based chemotherapy, or subjects in progression of disease after a maximum of one line of platinum-based therapy for advanced disease.
* Disease not amenable to curative surgery.
* Measurable disease, per modified Response Evaluation Criteria in Solid Tumor [RECIST] for pleural mesothelioma or RECIST version 1.1 for peritoneal mesothelioma).
* Life expectancy ≥ 12 weeks.
* ECOG performance status of 0 or 1
* Normal laboratory tests
* Negative screening tests for HIV, Hepatitis B, and Hepatitis C.
* Availability of archival tumor tissue or feasibility to perform a new tumor biopsy at screening phase.
* Men and women, of and over 18 years old. Women of childbearing potential (WOCBP) must use appropriate method(s) of contraception. WOCBP should use an adequate method to avoid pregnancy for 180 days after the last dose of investigational drug.

Exclusion Criteria:

* Involvement in the planning and/or conduct of the study.
* Participation in another clinical study with an investigational product during the last 6 weeks.
* Any previous treatment with a CTLA4, PD-1 or PD-L1 inhibitor, including tremelimumab or MEDI4736.
* History of another primary malignancy except for: malignancy treated with curative intent and with no known active disease ≥3 years before the first dose of study drug and of low potential risk for recurrence. Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease. Adequately treated carcinoma in situ without evidence of disease eg, cervical cancer in situ.
* Receipt of the last dose of anti-cancer therapy ≤ 6 weeks prior to the first dose of study drug.
* Mean QT interval corrected for heart rate (QTc) ≥470 ms using Bazett's Correction.
* Current or prior use of immunosuppressive medication within 28 days before the first dose of tremelimumab and MEDI4736, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid.
* Any unresolved toxicity (CTCAE grade >2) from previous anti-cancer therapy.
* Any prior Grade >3 immune-related adverse event (irAE) while receiving any previous immunotherapy agent, or any unresolved irAE >Grade 1. Active or prior documented autoimmune or inflammatory disorders
* History of primary immunodeficiency or allogeneic organ transplant.
* History of hypersensitivity to tremelimumab or MEDI4736 or any excipient.
* Uncontrolled intercurrent illness including, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, active peptic ulcer disease or gastritis, active bleeding diatheses
* Known history of previous clinical diagnosis of tuberculosis.
* History of leptomeningeal carcinomatosis.
* Receipt of live attenuated vaccination within 30 days prior to study entry or within 30 days of receiving tremelimumab and MEDI4736.
* Symptomatic or uncontrolled brain metastases requiring concurrent treatment, inclusive of but not limited to surgery, radiation and/or corticosteroids.
* Subjects with uncontrolled seizures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-06 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
immune-related (ir)- objective response rate (ORR) | 60 weeks
  proportion of subjects with complete response [CR] or partial Response [PR]) according to the ir-modified-RECIST or ir-RECIST 1.1 in pleural or peritoneal subjects, respectively.

SECONDARY OUTCOMES:
Immune-related-Disease control rate (ir-DCR) | 60 weeks
  proportion of subjects with ir-CR, ir-PR, ir-stable disease according to the ir-modified-RECIST or ir-RECIST 1.1 in pleural or peritoneal subjects, respectively
Disease control rate (DCR) | 60 weeks
  proportion of subjects with CR, PR, stable disease according to the modified-RECIST or RECIST 1.1 in pleural or peritoneal subjects, respectively
Immune-related-progression-free-survival (PFS) | 60 weeks
  ir-PFS per ir-modified-RECIST or ir-RECIST-1.1 for pleural or peritoneal mesothelioma respectively, will be defined as the time between the date of randomization and the date of progression or death
progression-free-survival (PFS) | 60 weeks
  PFS per modified-RECIST or RECIST-1.1 for pleural or peritoneal mesothelioma respectively, will be defined as the time between the date of randomization and the date of progression or death
Overall survival (OS) | 120 weeks
  Overall Survival (OS) is defined as the time from randomization until the date of death. For those subjects who have not died, OS will be censored at the recorded last date of subject contact, and for subjects with a missing recorded last date of contact, OS will be censored at the last date the subject was known to be alive.
Safety (adverse events) | 120 weeks
  The safety endpoints include adverse events (AEs) and serious adverse events (SAEs). Reporting of safety, extent of exposure, concomitant medications and discontinuation of study therapy will be based on all subjects who received at least 1 dose of treatment. Toxicity will be registered according to the NCICTC v 4.0
Immune-related-ORR based on PD-L1 tumor expression | 60 weeks
  proportion of subjects with PD-L1 positive or negative tumor expression who achieved a complete response [CR] or partial Response [PR]) according to the ir-modified-RECIST or ir-RECIST 1.1 in pleural or peritoneal subjects, respectively.
Immune-related-Disease control rate based on PD-L1 tumor expression | 60 weeks
  proportion of subjects with PD-L1 positive or negative tumor expression who achieved a CR, PR, stable disease according to the ir-modified-RECIST or ir-RECIST 1.1 in pleural or peritoneal subjects, respectively
Immune-related-progression- free-survival based on PD-L1 tumor expression | 60 weeks
  ir-PFS per ir-modified-RECIST or ir-RECIST-1.1 for pleural or peritoneal mesothelioma respectively, will be defined in subjects with PD-L1 positive or negative tumor expression as the time between the date of randomization and the date of progression or death
Overall survival based on PD-L1 tumor expression | 120 weeks
  Overall Survival (OS) is defined in subjects with PD-L1 positive or negative tumor expression as the time from randomization until the date of death. For those subjects who have not died, OS will be censored at the recorded last date of subject contact, and for subjects with a missing recorded last date of contact, OS will be censored at the last date the subject was known to be alive.

CONTACTS AND LOCATIONS:
Overall Officials: Luana Calabro', MD, PhD, Principal Investigator — Medical Oncology and Immunotherapy Division, Univeristy Hospital os Siena, Siena, Italy
Locations (1):
- Medical Oncology and Immunotherapy Division, University Hospital of Siena, Siena, Italy

REFERENCES:
- [Background] Calabro L, Morra A, Fonsatti E, Cutaia O, Amato G, Giannarelli D, Di Giacomo AM, Danielli R, Altomonte M, Mutti L, Maio M. Tremelimumab for patients with chemotherapy-resistant advanced malignant mesothelioma: an open-label, single-arm, phase 2 trial. Lancet Oncol. 2013 Oct;14(11):1104-1111. doi: 10.1016/S1470-2045(13)70381-4. Epub 2013 Sep 11. PMID 24035405
- [Background] Calabro L, Ceresoli GL, di Pietro A, Cutaia O, Morra A, Ibrahim R, Maio M. CTLA4 blockade in mesothelioma: finally a competing strategy over cytotoxic/target therapy? Cancer Immunol Immunother. 2015 Jan;64(1):105-12. doi: 10.1007/s00262-014-1609-9. Epub 2014 Sep 19. PMID 25233793
- [Background] Calabro L, Morra A, Fonsatti E, Cutaia O, Fazio C, Annesi D, Lenoci M, Amato G, Danielli R, Altomonte M, Giannarelli D, Di Giacomo AM, Maio M. Efficacy and safety of an intensified schedule of tremelimumab for chemotherapy-resistant malignant mesothelioma: an open-label, single-arm, phase 2 study. Lancet Respir Med. 2015 Apr;3(4):301-9. doi: 10.1016/S2213-2600(15)00092-2. Epub 2015 Mar 26. PMID 25819643
- [Background] Antonia et al. A Phase Ib study of MEDI4736, a programmed cell death ligand-1 (PD-L1) antibody, in combination with tremelimumab, a cytotoxic T-lymphocyte-associated protein-4 (CTLA-4) antibody, in patients with advanced non-small cell lung cancer (NSCLC). ASCO 2015 (Abstract #3014).
- [Derived] Calabro L, Rossi G, Morra A, Rosati C, Cutaia O, Daffina MG, Altomonte M, Di Giacomo AM, Casula M, Fazio C, Palmieri G, Giannarelli D, Covre A, Maio M. Tremelimumab plus durvalumab retreatment and 4-year outcomes in patients with mesothelioma: a follow-up of the open label, non-randomised, phase 2 NIBIT-MESO-1 study. Lancet Respir Med. 2021 Sep;9(9):969-976. doi: 10.1016/S2213-2600(21)00043-6. Epub 2021 Apr 9. PMID 33844995
- [Derived] Calabro L, Morra A, Giannarelli D, Amato G, D'Incecco A, Covre A, Lewis A, Rebelatto MC, Danielli R, Altomonte M, Di Giacomo AM, Maio M. Tremelimumab combined with durvalumab in patients with mesothelioma (NIBIT-MESO-1): an open-label, non-randomised, phase 2 study. Lancet Respir Med. 2018 Jun;6(6):451-460. doi: 10.1016/S2213-2600(18)30151-6. Epub 2018 May 15. PMID 29773326
- See also: Fondazione NIBIT — http://www.fondazionenibit.org/